CLINICAL TRIAL: NCT02391883
Title: Hip-Fracture Surgery on Patients in Clopidogrel Therapy
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Peter Toft Tengberg, Consultant, Hvidovre University Hospital
Other Study IDs: CLOP-HIPFX study
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Hip Fracture
Keywords: clopidogrel therapy; platelet aggregation inhibitor; adverse event
MeSH Terms: conditions — Hip Fractures | interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Clopidogrel: Patients in Clopidogrel or Dual Antiplatelet Therapy (Clopidogrel+Acetylsalicylic acid) at the time of admission AND who are operated <24 hours after admission.
  Interventions: Drug: Clopidogrel
- Control: Patients NOT in anticoagulation treatment (Except acetylsalicylic acid) AND who are operated <24 hours after admission.

INTERVENTIONS:
Drug: Clopidogrel
  Groups: Clopidogrel

SUMMARY:
Patients in Clopidogrel therapy alone or in combination with acetylsalicylic acid (Dual Antiplatelet Therapy (DAPT) presenting with a hip-fracture represent the surgeon with the dilemma of putting the patient at risk of a major blood loss during and after surgery, or putting the patient at risk of a thromboembolic event after surgery. The investigators hypothesize that the risk of a major blood loss in patients that are still under the effect of Clopidogrel or DAPT during or after hip-fracture surgery is relatively low. The investigators have conducted a retrospective observational study on hip-fracture patients to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* All patients operated with short intramedullary nail for hip-fractures, in the study period. (1st of Jan. 2011-31st of Dec. 2013)

Exclusion Criteria:

* patients operated >24 hours after admission, patients in other forms of anticoagulation medication except acetylsalicylic acid (including vitamin K antagonists, dipyridamole, dabigatran, apixaban and rivaroxaban), missing data on blood loss in patient chart, missing blood samples in the first 4 days and extra-national patients (follow up not possible). Patients operated on both sides during the inclusion period were only included with data on their latest operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 356 patients were included in the final analysis. Out of this group we identified 36 patients taking Clopidogrel. 24 of these were in DAPT. 12 patients were in Clopidogrel therapy alone. The indications for treatment were: CNS thrombosis (n=14); Unstable Angina (n=8); Peripheral Atherosclerosis (n=3); Myocardial Infarction (n=2); Insertion of stent >24 months earlier (n=1); and Unknown indication (n=8). All patients had their treatment discontinued on admission.
  All analyzed patients were operated within 24 hours of admission (n=356).
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Surgical Blood Loss | at time of surgery
  Blood loss as assessed by the surgeon

SECONDARY OUTCOMES:
Total BLood Loss | From admission to third day after surgery.
  Calculated based on the method described by Foss et al 2006 (Hidden Blood Loss in hip fractures)
Number of transfusions | From admission to third day after surgery
  Number of Red Blood Cell transfusions
30 and 90 day mortality | 30 and 90 days postoperatively
  Recorded from national persons registry (CPR-registeret)
Massive transfusion | within 24 hours of surgery
  >10 Red Blood Cell transfusion within 24 hours of surgery.